CLINICAL TRIAL: NCT02711878
Title: Healing Hearts and Mending Minds in Older Adults Living With HIV
Acronym: FitBrain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Drenna Waldrop-Valverde, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00080302; 1R01NR014973-01 (NIH)
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Results first posted 2022-07-01 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: HIV; Cardiovascular Disease; AIDS
MeSH Terms: conditions — Cardiovascular Diseases; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Let's Move Program (Experimental): Participants in this group will be asked to walk five times per week for twelve weeks for a minimum of 30 minutes in their home while wearing a heart rate monitor and a pedometer. Participants will then enter a maintenance exercise period for 65 weeks.
  Interventions: Behavioral: Let's Move Program; Behavioral: Group Motivational Interviewing
- Let's Flex Program (Active Comparator): Participants in this group will be asked to stretch five times per week for twelve weeks for a minimum of thirty minutes in their home. Participants will then enter a maintenance exercise period for 65 weeks.
  Interventions: Behavioral: Let's Flex Program; Behavioral: Group Motivational Interviewing

INTERVENTIONS:
Behavioral: Let's Move Program — Participants will be asked to walk five times per week for twelve weeks for a minimum of 30 minutes while wearing a heart rate monitor and a pedometer. Participants will also receive weekly telephone calls from a member of the research team to monitor walking progress and to change walking duration or intensity level based on their progress.After the twelve week period, participants will enter a maintenance exercise phase for weeks 13-17 in which they will be asked to maintain their exercise regimen.
  Arms: Let's Move Program
Behavioral: Let's Flex Program — Participants will be asked to stretch five times per week for twelve weeks for a minimum of 30 minutes. Participants will also receive weekly telephone calls from a member of the research team to monitor progress and to change duration or intensity level based on their progress.After the twelve week period, participants will enter a maintenance exercise phase for weeks 13-17 in which they will be asked to maintain their exercise regimen.
  Arms: Let's Flex Program
Behavioral: Group Motivational Interviewing — Participants will attend four separate group intervention sessions for 2.5 hours for four consecutive weeks at the beginning of the program. Groups will consist of 6-8 members and will focus on the rationale for aerobic exercise, barriers to exercise, finding time for exercise, how to set short and long term exercise goals, and use of self-monitoring to improve exercise engagement.

SUMMARY:
The purpose of this study is to see if exercise is helpful for improving memory, concentration thinking abilities, physical function, and quality of life for adults aged 50 to 89 years living with HIV and who have two or more cardiovascular disease risk factors. The study will test two kinds of intervention exercises: one group will walk for exercise and the second group will stretch for exercise. Members of both interventions will be asked to participate in one-on-one interviews/assessments, measures of physical functioning, and some sessions with others who are also enrolled in the study.

DETAILED DESCRIPTION:
This is a two arm, randomized controlled trial to test the longitudinal effects of the Let's Move Program (walking for exercise) compared to effects of the attention control Let's Flex Program (stretching for exercise) in participants aged 50 to 89 years living with HIV and who have two or more cardiovascular disease risk factors. Participants in both interventions will be asked to participate in one-on-one interviews/assessments, measures of physical functioning, and some sessions with others who are also enrolled in the study. Participants will participate in an in home exercise program for twelve weeks in which the study team will help identify maximum duration and intensity followed by a maintenance period for weeks 13-58.

ELIGIBILITY:
Inclusion Criteria:

* HIV diagnosis
* English speaking
* Live independently within a 30-45 mile radius of Atlanta, Georgia
* Not involved in any structured exercise program or exercising 3 or more times per week for a minimum of 30 minutes
* Not involved in any weight loss program
* Not hospitalized within the last 60-days
* Clinically stable and on antiretroviral therapy (ART) 6 months before enrollment
* If taking statins, stable on medication for 3 months
* Score 3 or less on the verbal memory subtest of the Montreal Cognitive Assessment (MoCA)
* Less than 0.5 standard deviations (SD) below mean on the Oral Trail Making Test B
* Able to provide informed consent and pass a consent post-test

Exclusion Criteria:

* Non sedentary (defined as engaging in > 30 minutes of moderately strenuous exercise 3 times or more a week)
* Medical or physical condition that would preclude participation in the exercise component of the study (e.g., severe arthritis or mobility problems, lower extremity amputations, joint replacement(s), balance disorders, dizziness, dyspnea on exertion (DOE) with moderate exertion, difficulty walking one block, recent falls, obvious injury to lower extremity, uncontrolled hypertension or diabetes, renal failure, blindness, or a history of angina with activity)
* Ischemic changes or inappropriate BP changes on baseline exercise (modified Balke or Bruce) treadmill test
* On oral corticosteroids (nasal, optical and inhaler corticosteroids allowed without restriction) , experiencing acute inflammation at time of baseline or follow-up testing (this will result in rescheduling of testing if no other exclusion criteria apply after 2 weeks)
* Presence of current opportunistic infection
* Any terminal illness
* Regular use of anti-inflammatory medications such as non-steroidal anti-inflammatory agents excluding low dose aspirin
* On anti-psychotics
* On tricyclic antidepressants
* On anti-depressants equal to the equivalent of more than 1 mg of Clonazepam
* On Lithium
* Women who are pregnant
* Severe learning disabilities, intellectual disabilities, schizophrenia, bipolar, psychotic disorders to minimize confounding effects on neurocognitive data
* Confounding neuro-medical conditions (e.g., active central nervous system (CNS) opportunistic infections, seizure disorders, head injury with loss of consciousness greater than 30 minutes, intracranial neoplasms, stroke with neurological or neuropsychiatric sequelae, and non-HIV-associated dementias)
* Meet criteria for any Substance Use Disorder or Major Depression within 6 months of evaluation
* Creatinine > 2.5 within the past 6 months
* Patient Health Questionnaire-2 (PHQ-2) score > 4
* Completed 8 years or less of school
* Failed to pass post-consent test after three attempts
* Two or more positive drug screen tests
* Alcohol breathalyzer test result > 0.03

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2016-09; Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Drenna Waldrop-Valverde, PhD, Principal Investigator — Emory University; Rebecca Gary, PhD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Ponce De Leon Center, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between September 2016 and December 2018.
Period: Overall Study
Arm/Group | Let's Move Program | Let's Flex Program
Started | 76 | 39
Completed Visit T1 (13-15 Weeks Post Baseline) | 69 | 33
Completed Visit T2 (28-30 Weeks Post Baseline) | 68 | 33
Completed Visit T3 (56-58 Weeks Post Baseline) | 72 | 31
Completed | 68 | 33
Not Completed | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Let's Move Program | Let's Flex Program | Total
Number analyzed (Participants) | 76 | 39 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 73 | 38 | 111
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.68 (5.2) | 53.92 (5.2) | 55.09 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 20 | 46
  Male | 50 | 19 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 63 | 37 | 100
  White | 10 | 2 | 12
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants] — Data was collected at the School of Nursing and at the Clinical Translational Science Institute of Atlanta at each measurement point.
  Participants
    United States | 76 | 39 | 115

OUTCOME MEASURES:

1. Primary Outcome: Stroop Color and Word Test Score
Description: The Stroop Color and Word Test is a performance-based test of executive function and inhibitory responding. The participant is presented with a page with the words "red, blue, and green" printed 100 times in (20 words in 5 columns). Each word is printed in a different color of ink than the target word (e.g, the word "red" is printed in blue ink). Participants read the color of ink in which the word is printed as quickly are possible within a time limit. The correct number within the time limit is the score. Raw scores (unadjusted for age and education) range from 0-100.
Time Frame: Baseline, T1 (13-15 weeks post baseline), T2 (28-30 weeks post baseline), T3 ( 56-58 weeks post baseline)
Population: The number analyzed includes participants who were able to complete each study visit.
Measure: Mean (Standard Deviation); unit: number of correct responses
Arm/Group | Let's Move Program | Let's Flex Program
Number analyzed (Participants) | 76 | 39
number of correct responses
  Baseline | 31.17 (8.13) | 28.89 (7.59)
  T1 (13-15 weeks post baseline): number analyzed (Participants) | 69 | 33
  T1 (13-15 weeks post baseline) | 32.87 (8.85) | 30.69 (6.64)
  T2 (28-30 weeks post baseline): number analyzed (Participants) | 68 | 33
  T2 (28-30 weeks post baseline) | 33.09 (8.72) | 30.39 (9.5)
  T3 ( 56-58 weeks post baseline): number analyzed (Participants) | 72 | 31
  T3 ( 56-58 weeks post baseline) | 33.44 (8.74) | 31.77 (7.83)

2. Primary Outcome: Trail Making Test Score
Description: The Trail Making Test is a performance based test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect circles as possible while still maintaining accuracy. Trails A subtest requires the connection in sequence of 25 circles labeled by numbers. Trails B requires the connection in sequence of 25 circles labeled by alternating numbers and letters (1-A-2-B-3-C). The score on the test is the time in seconds that it takes to complete.
  Higher scores (i.e., time) indicate poorer performance.
Time Frame: Baseline, T1 (13-15 weeks post baseline), T2 (28-30 weeks post baseline), T3 ( 56-58 weeks post baseline)
Population: The number analyzed includes participants who were able to complete each study visit.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Let's Move Program | Let's Flex Program
Number analyzed (Participants) | 76 | 39
seconds
  Part A - Baseline | 35.84 (14.11) | 37.74 (20.08)
  Part A -T1 (13-15 weeks post baseline): number analyzed (Participants) | 69 | 33
  Part A -T1 (13-15 weeks post baseline) | 33.62 (12.39) | 35.58 (16.51)
  Part A - T2 (28-30 weeks post baseline): number analyzed (Participants) | 68 | 33
  Part A - T2 (28-30 weeks post baseline) | 34.73 (17.54) | 39.03 (15.62)
  Part A - T3 ( 56-58 weeks post baseline): number analyzed (Participants) | 72 | 31
  Part A - T3 ( 56-58 weeks post baseline) | 33.29 (12.49) | 36.23 (12.92)
  Part B - Baseline | 113.7 (62.29) | 137.95 (86.58)
  Part B -T1 (13-15 weeks post baseline): number analyzed (Participants) | 69 | 33
  Part B -T1 (13-15 weeks post baseline) | 109.51 (58.68) | 142.26 (93.74)
  Part B - T2 (28-30 weeks post baseline): number analyzed (Participants) | 68 | 33
  Part B - T2 (28-30 weeks post baseline) | 117.91 (82.97) | 164.58 (128.75)
  Part B - T3 ( 56-58 weeks post baseline): number analyzed (Participants) | 72 | 31
  Part B - T3 ( 56-58 weeks post baseline) | 115.76 (94.08) | 145.28 (115.38)

3. Primary Outcome: Letter Fluency Assessed by Change in FAS Test Score
Description: The FAS test requires stating out loud as many words that begin with the assigned letter (F, A, and S) as possible within 60-seconds. Results represent total number of words stated for F,A & S combined.
Time Frame: Baseline, T1 (13-15 weeks post baseline), T2 (28-30 weeks post baseline), T3 ( 56-58 weeks post baseline)
Population: The number analyzed includes participants who were able to complete each study visit.
Measure: Mean (Standard Deviation); unit: number of correct words
Arm/Group | Let's Move Program | Let's Flex Program
Number analyzed (Participants) | 76 | 39
number of correct words
  Baseline | 35.91 (10.67) | 31.44 (8.64)
  T1 ( 13-15 weeks post baseline): number analyzed (Participants) | 69 | 33
  T1 ( 13-15 weeks post baseline) | 38.51 (11.48) | 31.28 (9.1)
  T2 (28-30 weeks post baseline): number analyzed (Participants) | 68 | 33
  T2 (28-30 weeks post baseline) | 37.26 (11.18) | 34.33 (11.01)
  T3 ( 56-58 weeks post baseline): number analyzed (Participants) | 72 | 31
  T3 ( 56-58 weeks post baseline) | 38.24 (11.93) | 35.4 (13.96)

4. Primary Outcome: Category Fluency Test Score
Description: The category fluency test requires participants to state out load the names of as many animals as possible within 60-seconds. Results are total number of animals named.
Time Frame: Baseline, T1 (13-15 weeks post baseline), T2 (28-30 weeks post baseline), T3 ( 56-58 weeks post baseline)
Population: Some participants did not complete the form or completed the incorrect forms and could not be included in the analysis.
Measure: Mean (Standard Deviation); unit: Number of correct animals named
Arm/Group | Let's Move Program | Let's Flex Program
Number analyzed (Participants) | 76 | 39
Number of correct animals named
  Baseline | 19.97 (4.96) | 18.89 (6.03)
  T1 (13-15 weeks post baseline): number analyzed (Participants) | 69 | 33
  T1 (13-15 weeks post baseline) | 19.87 (4.35) | 17.63 (6.59)
  T2 (28-30 weeks post baseline): number analyzed (Participants) | 68 | 33
  T2 (28-30 weeks post baseline) | 20.24 (4.38) | 17.82 (6.26)
  T3 (56-58 weeks post baseline): number analyzed (Participants) | 72 | 31
  T3 (56-58 weeks post baseline) | 19.22 (4.7) | 17.13 (5.53)

5. Primary Outcome: Hopkins Verbal Learning Test (HVLT) - Revised Score
Description: The HVLT-Revised is a list learning task requiring the respondent to recall as many words as possible from a list of 12 words provided orally by the examiner. There is a learning trial, a delayed recall trial, and a recognition trial. Results show HVLT Total recall (Total number if words recalled over 3 trials) and HVLT Delayed recall (Total number of words recalled after 25 minute delay).
Time Frame: Baseline, T1 (13-15 weeks post baseline), T2 (28-30 weeks post baseline), T3 ( 56-58 weeks post baseline)
Population: Some participants did not complete the form or completed the incorrect forms and could not be included in the analysis.
Measure: Mean (Standard Deviation); unit: Number of correct words recalled
Arm/Group | Let's Move Program | Let's Flex Program
Number analyzed (Participants) | 75 | 39
Number of correct words recalled
  Total recall - Baseline | 6.65 (2.57) | 6.46 (2.4)
  Total recall - T1 ( 13-15 weeks post baseline): number analyzed (Participants) | 68 | 39
  Total recall - T1 ( 13-15 weeks post baseline) | 6.87 (2.37) | 6.65 (2.17)
  Total recall - T2 (28-30 weeks post baseline): number analyzed (Participants) | 68 | 39
  Total recall - T2 (28-30 weeks post baseline) | 6.56 (2.68) | 7 (2.25)
  Total recall - T3 ( 56-58 weeks post baseline): number analyzed (Participants) | 72 | 31
  Total recall - T3 ( 56-58 weeks post baseline) | 5.93 (2.6) | 6.35 (2.68)
  Delayed recall - Baseline: number analyzed (Participants) | 74 | 39
  Delayed recall - Baseline | 6.65 (2.57) | 6.46 (2.4)
  Delayed recall - T1 ( 13-15 weeks post baseline): number analyzed (Participants) | 68 | 33
  Delayed recall - T1 ( 13-15 weeks post baseline) | 6.87 (2.37) | 6.65 (2.17)
  Delayed recall - T2 (28-30 weeks post baseline): number analyzed (Participants) | 67 | 33
  Delayed recall - T2 (28-30 weeks post baseline) | 6.56 (2.68) | 7 (2.25)
  Delayed recall - T3 ( 56-58 weeks post baseline): number analyzed (Participants) | 72 | 31
  Delayed recall - T3 ( 56-58 weeks post baseline) | 5.93 (2.6) | 6.35 (2.68)

6. Primary Outcome: Brief Visual Memory Test - Revised (BVMT-R) Score
Description: The Brief Visual Memory Test is a performance based test that requires that participants reproduce simple visual images from memory (the images are displayed for 10 seconds then removed from view). The BVMT-R contains a learning trial, a recall trial, a recognition trial, and a copy trial. Each figure recalled is given 0,1, or 2 points based on accuracy and location recall. Results show BVMT Total recall (Total number if figures recalled over 3 trials: range 0 - 36) and BVMT delayed recall (total number of figures recalled after 25 min delay. Score range 0-12). Higher score correlate with better outcome.
Time Frame: Baseline, T1 (13-15 weeks post baseline), T2 (28-30 weeks post baseline), T3 ( 56-58 weeks post baseline)
Population: Some participants did not complete the form or completed the incorrect forms and could not be included in the analysis.
Measure: Mean (Standard Deviation); unit: number of correct figures recalled
Arm/Group | Let's Move Program | Let's Flex Program
Number analyzed (Participants) | 76 | 39
number of correct figures recalled
  Total recall - Baseline | 16.97 (7.02) | 15.97 (4.2)
  Total recall - T1 ( 13-15 weeks post baseline): number analyzed (Participants) | 69 | 33
  Total recall - T1 ( 13-15 weeks post baseline) | 19.99 (5.96) | 17.16 (4.59)
  Total recall - T2 (28-30 weeks post baseline): number analyzed (Participants) | 68 | 33
  Total recall - T2 (28-30 weeks post baseline) | 19.59 (6.78) | 18.18 (5.69)
  Total recall - T3 ( 56-58 weeks post baseline): number analyzed (Participants) | 72 | 31
  Total recall - T3 ( 56-58 weeks post baseline) | 17.47 (7.17) | 16.23 (7.36)
  Delayed recall - Baseline | 6.88 (2.84) | 6.51 (2.58)
  Delayed recall - T1 ( 13-15 weeks post baseline): number analyzed (Participants) | 69 | 33
  Delayed recall - T1 ( 13-15 weeks post baseline) | 7.59 (2.42) | 6.77 (2.03)
  Delayed recall - T2 (28-30 weeks post baseline): number analyzed (Participants) | 68 | 33
  Delayed recall - T2 (28-30 weeks post baseline) | 7.84 (2.81) | 7.67 (2.79)
  Delayed recall - T3 ( 56-58 weeks post baseline): number analyzed (Participants) | 72 | 31
  Delayed recall - T3 ( 56-58 weeks post baseline) | 7.01 (2.88) | 6.29 (3.25)

7. Primary Outcome: Grooved Pegboard Test Score
Description: The Grooved Pegboard Test requires the placing of grooved pegs into a same-shaped hole as quickly as possible, once with the dominant hand and once with the non-dominant hand.
Time Frame: Baseline, T1 (13-15 weeks post baseline), T2 (28-30 weeks post baseline), T3 ( 56-58 weeks post baseline)
Population: The number analyzed includes participants who were able to complete each study visit.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Let's Move Program | Let's Flex Program
Number analyzed (Participants) | 76 | 39
Seconds
  Dominant Hand - Baseline | 100.26 (52.08) | 103.46 (44.52)
  Dominant Hand - T1 ( 13-15 weeks post baseline): number analyzed (Participants) | 69 | 33
  Dominant Hand - T1 ( 13-15 weeks post baseline) | 91.49 (26.16) | 101.94 (30.38)
  Dominant Hand -T2 (28-30 weeks post baseline): number analyzed (Participants) | 68 | 33
  Dominant Hand -T2 (28-30 weeks post baseline) | 90.81 (32.85) | 101.78 (35.76)
  Dominant Hand -T3 (56-58 weeks post baseline): number analyzed (Participants) | 72 | 31
  Dominant Hand -T3 (56-58 weeks post baseline) | 89.99 (34.03) | 92.45 (29.37)
  Nondominant Hand - Baseline: number analyzed (Participants) | 76 | 33
  Nondominant Hand - Baseline | 111.97 (48.88) | 118.67 (56.29)
  Nondominant Hand - T1 ( 13-15 weeks post baseline): number analyzed (Participants) | 69 | 33
  Nondominant Hand - T1 ( 13-15 weeks post baseline) | 110.63 (43.35) | 120.42 (37.18)
  Nondominant Hand -T2 (28-30 weeks post baseline): number analyzed (Participants) | 68 | 33
  Nondominant Hand -T2 (28-30 weeks post baseline) | 108.75 (50.43) | 119.06 (43.12)
  Nondominant Hand -T3 (56-58 weeks post baseline): number analyzed (Participants) | 72 | 31
  Nondominant Hand -T3 (56-58 weeks post baseline) | 101.04 (46.31) | 112.5 (41.98)

8. Primary Outcome: Finger Tapping Test Score
Description: The finger tapping test a fine motor speed requires tapping a lever with the index finger as quickly as possible. Trials with the dominant and non-dominant hand are completed.
Time Frame: Baseline, T1 (13-15 weeks post baseline), T2 (28-30 weeks post baseline), T3 ( 56-58 weeks post baseline)
Population: The number analyzed includes participants who were able to complete each study visit.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Let's Move Program | Let's Flex Program
Number analyzed (Participants) | 76 | 39
Seconds
  Dominant hand - Baseline | 36.21 (8.13) | 32.83 (9.89)
  Dominant hand -T1 ( 13-15 weeks post baseline): number analyzed (Participants) | 69 | 33
  Dominant hand -T1 ( 13-15 weeks post baseline) | 39.34 (10.47) | 33.9 (11.37)
  Dominant hand -T2 ( 28-30 weeks post baseline): number analyzed (Participants) | 68 | 33
  Dominant hand -T2 ( 28-30 weeks post baseline) | 38.19 (8.98) | 34.31 (8.72)
  Dominant hand -T2 ( 56-58 weeks post baseline): number analyzed (Participants) | 72 | 31
  Dominant hand -T2 ( 56-58 weeks post baseline) | 38.82 (9.57) | 33.13 (6.92)
  Nondominant hand - Baseline | 34.85 (8.29) | 33.29 (10.09)
  Nondominant hand -T1 ( 13-15 weeks post baseline): number analyzed (Participants) | 69 | 33
  Nondominant hand -T1 ( 13-15 weeks post baseline) | 36.59 (8.32) | 33.98 (9.51)
  Nondominant hand -T2 ( 28-30 weeks post baseline): number analyzed (Participants) | 68 | 33
  Nondominant hand -T2 ( 28-30 weeks post baseline) | 35.94 (8.05) | 34.53 (11.61)
  Nondominant hand -T2 ( 56-58 weeks post baseline): number analyzed (Participants) | 71 | 31
  Nondominant hand -T2 ( 56-58 weeks post baseline) | 36.91 (8.36) | 31.94 (7.39)

9. Primary Outcome: Coding Test Score
Description: The coding test requires writing the corresponding symbol associated with a letter from a key provided. As many responses as possible are completed in the 120 second time limit. Results presented are the total number of correct responses (possible score range 0-135).
Time Frame: Baseline, T1 (13-15 weeks post baseline), T2 (28-30 weeks post baseline), T3 ( 56-58 weeks post baseline)
Population: The number analyzed includes participants who were able to complete each study visit.
Measure: Mean (Standard Deviation); unit: number of correct responses
Arm/Group | Let's Move Program | Let's Flex Program
Number analyzed (Participants) | 76 | 39
number of correct responses
  Baseline | 46.07 (14.64) | 45.69 (15.44)
  T1 (13-15 weeks post baseline): number analyzed (Participants) | 69 | 33
  T1 (13-15 weeks post baseline) | 45.31 (16.14) | 43.13 (14.58)
  T2 (28-30 weeks post baseline): number analyzed (Participants) | 68 | 33
  T2 (28-30 weeks post baseline) | 47.89 (17.32) | 42.84 (15.19)
  T3 (56-58 weeks post baseline): number analyzed (Participants) | 72 | 31
  T3 (56-58 weeks post baseline) | 50.11 (16.41) | 47.23 (14.93)

10. Primary Outcome: Digit Span Test Score
Description: The digit span test is a performance based test that requires repeating an increasing span of digits that are provided verbally by the examiner. The test includes trials of repeating digits in the same order presented by the examiner, in the reverse order of that presented by the examiner, and in ascending sequence. Scores range from 0 to 48. Higher score correlates with better outcome.
Time Frame: Baseline, T1 (13-15 weeks post baseline), T2 (28-30 weeks post baseline), T3 ( 56-58 weeks post baseline)
Population: The number analyzed includes participants who were able to complete each study visit.
Measure: Mean (Standard Deviation); unit: number of correct digits
Arm/Group | Let's Move Program | Let's Flex Program
Number analyzed (Participants) | 79 | 39
number of correct digits
  Baseline | 23.19 (5.63) | 21.67 (5.56)
  T1 (13-15 weeks post baseline): number analyzed (Participants) | 69 | 33
  T1 (13-15 weeks post baseline) | 24.32 (5.16) | 22.41 (4.72)
  T2 (28-30 weeks post baseline): number analyzed (Participants) | 68 | 33
  T2 (28-30 weeks post baseline) | 23.86 (6.62) | 21.76 (5.84)
  T3 ( 56-58 weeks post baseline): number analyzed (Participants) | 71 | 31
  T3 ( 56-58 weeks post baseline) | 23.86 (6.32) | 21.27 (5.56)

11. Primary Outcome: Symbol Span Test Score
Description: The subtest assesses visual working memory using novel visual stimuli. A series of abstract symbols on a page are shown briefly. Then the symbols are to be selected from an array of symbols in the same order they were presented on the previous page. This performance based test measures storage and manipulation of visual details in working memory. Score range from 0-36. Higher score correlates with better outcome.
Time Frame: Baseline, 3 months, 6 months and 12 months Post Intervention
Population: The number analyzed includes participants who were able to complete each study visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Let's Move Program | Let's Flex Program
Number analyzed (Participants) | 76 | 39
score on a scale
  Baseline | 17.19 (6.11) | 15.33 (5.89)
  3 months post-intervention: number analyzed (Participants) | 69 | 32
  3 months post-intervention | 19.56 (5.76) | 16.78 (5.58)
  6 months post-intervention: number analyzed (Participants) | 68 | 33
  6 months post-intervention | 19.17 (7.16) | 17.18 (6.38)
  12 months post-intervention: number analyzed (Participants) | 72 | 32
  12 months post-intervention | 19.56 (5.76) | 16.78 (5.58)

12. Primary Outcome: Instrumental Activities of Daily Living (IADL) Test Score
Description: The Instrumental Activities of Daily Living (IADL) Test is a self-report measure assessing the amount of assistance, if any, required to do day-to-day tasks necessary to live independently. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women and 0 through 5 for men to avoid potential gender bias). Higher scores indicate worse performance in instrumental activities activities of daily living.
Time Frame: Baseline, T1 (13-15 weeks post baseline), T2 (28-30 weeks post baseline), T3 (56-58 weeks post baseline)
Population: The number analyzed includes participants who were able to complete each study visit.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Let's Move Program | Let's Flex Program
Number analyzed (Participants) | 74 | 38
Score on a scale
  Baseline | 7.95 (0.19) | 7.86 (0.66)
  T1 (13-15 weeks post baseline): number analyzed (Participants) | 66 | 30
  T1 (13-15 weeks post baseline) | 7.96 (0.24) | 7.9 (0.30)
  T2 (28-30 weeks post baseline): number analyzed (Participants) | 62 | 30
  T2 (28-30 weeks post baseline) | 7.83 (0.65) | 7.93 (0.25)
  T3 (56-58 weeks post baseline): number analyzed (Participants) | 59 | 28
  T3 (56-58 weeks post baseline) | 7.89 (0.44) | 7.71 (0.76)

13. Primary Outcome: NIH Toolbox
Description: Computerized cognitive tests developed and distributed by the NIH. Tests include Pattern Comparison Processing Speed Test, Picture Vocabulary Test, Reading Recognition Test, Dimensional Change Card Sort Test, Flanker Inhibitory Control and Attention Test, Picture Sequence Memory Test, List Sorting Working Memory Test, and Oral Symbol Digit Test
Time Frame: Baseline, Post Intervention (Up to 58 weeks)
Population: In order to reduce participant burden, the NIH toolbox neurocognitive tests were not administered because was redundant with the outcomes measured by the other cognitive tests.
Arm/Group | Let's Move Program | Let's Flex Program
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Soluble Cluster of Differentiation 14 (sCD14) Level
Description: Soluble Cluster of Differentiation 14 (sCD14) is a marker of monocyte activation, is associated with neurocognitive impairment and HIV-associated neurocognitive disorders (HANDs) and higher mortality in persons living with HIV.
Time Frame: Baseline, T1 (13-15 weeks), T2 (28-30 weeks), T3 (56 -58 weeks)
Population: Lab assays were completed at each time-point based on the participants availability and those samples that were good for lab processing.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Let's Move Program | Let's Flex Program
Number analyzed (Participants) | 59 | 27
pg/ml
  Baseline | 2306.0 (711.94) | 2373.1 (525.3)
  T1 (13-15 weeks) | 2315.5 (748.5) | 2342.6 (672.5)

15. Secondary Outcome: Interleukin 6 (IL-6) Level
Description: IL-6 is a pro-inflammatory cytokine known to contribute to the pathogenesis of risk of cardiovascular disease (CVD) and cognitive impairment (CI) through inflammation and promotion of endothelial vascular dysfunction. IL-6 is measured by enzyme-linked immunosorbent assay (ELISA) and reported as in picograms per deciliter (pg/dL). Higher concentrations of IL-6 raise congenital heart defect risk.
Time Frame: Baseline, T1 (13-15 Weeks), T2 (28-30 weeks), T3 (56-58 weeks)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Let's Move Program | Let's Flex Program
Number analyzed (Participants) | 53 | 24
pg/ml
  Baseline | 2.5 (3.09) | 5.4 (12.5)
  T1 (13-15 wks) | 2.5 (3.2) | 5.1 (10.9)
  T2 (28-30 wks) | 2.3 (2.06) | 4.7 (9.9)
  T3 (56-58 wks) | 2.5 (2.4) | 7.2 (17.6)

16. Secondary Outcome: Tumor Necrosis Factor Alpha (TNF-alpha) Level
Description: TNFR1 membrane bound receptors that have been shown to bind TNF alpha. Activation of TNFR1 mediates the proinflammatory properties of TNF alpha.
Time Frame: Baseline, T1 (13-15 wks), T2 (28-30 wks), T3 (56-58 wks)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Let's Move: Let's Move Program: Participants will be asked to walk five times per week for twelve weeks for a minimum of 30 minutes while wearing a heart rate monitor and a pedometer. Participants will also receive weekly telephone calls from a member of the research team to monitor walking progress and to change walking duration or intensity level based on their progress.
  After the twelve-week period, participants will enter a maintenance exercise phase for weeks 13-17 in which they will be asked to maintain their exercise regimen.
  Group Motivational Interviewing: Participants will attend four separate group intervention sessions for 2.5 hours for four consecutive weeks at the beginning of the program. Groups will consist of 6-8 members and will focus on the rationale for aerobic exercise, barriers to exercise, finding time for exercise, how to set short and long term exercise goals, and use of self-monitoring to improve exercise engagement.
- Let's Flex: Let's Flex Program: Participants will be asked to stretch five times per week for twelve weeks for a minimum of 30 minutes. Participants will also receive weekly telephone calls from a member of the research team to monitor progress and to change duration or intensity level based on their progress. After the twelve week period, participants will enter a maintenance exercise phase for weeks 13-17 in which they will be asked to maintain their exercise regimen.
  Group Motivational Interviewing: Participants will attend four separate group intervention sessions for 2.5 hours for four consecutive weeks at the beginning of the program. Groups will consist of 6-8 members and will focus on the rationale for aerobic exercise, barriers to exercise, finding time for exercise, how to set short and long term exercise goals, and use of self-monitoring to improve exercise engagement.
Arm/Group | Let's Move | Let's Flex
Number analyzed (Participants) | 55 | 25
pg/ml
  Baseline | 1.6 (1.1) | 1.6 (0.6)
  T1 (13-15 wks) | 1.7 (1.08) | 1.71 (0.74)
  T2 (28-30 wks) | 1.6 (1.03) | 1.75 (0.86)
  T3 (56-58 wks) | 1.6 (0.82) | 1.71 (0.80)

17. Secondary Outcome: Brain-derived Neurotrophic Factor (BDNF) Level
Description: BDNF is a protein that occurs naturally in the hippocampus, cortex, and basal forebrain-areas vital to learning, memory, and higher thinking; an increase in BDNF in animal models and humans is thought to enhance neurogenesis. BDNF is reported as in picogram per milliliter (pg/mL).
Time Frame: Baseline, Post Intervention (Up to 58 weeks)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Let's Move Program | Let's Flex Program
Number analyzed (Participants) | 56 | 23
pg/mL
  Baseline | 2436.95 (2376.96) | 2910.17 (2571.53)
  T1 (13-15 weeks) | 3142.40 (3378.12) | 2963.97 (2678.83)
  T2 (28-30 weeks) | 3014.45 (3941.81) | 2895.28 (2316.84)
  T3 (56-58 weeks) | 2347.42 (2877.94) | 4877.86 (7766.09)

18. Secondary Outcome: Flow-Mediated Dilatation (FMD)
Description: Flow-mediated dilatation (FMD) is a measure of endothelial function; the measure of % FMD at 60 seconds reflects arterial relaxation time after cuff deflation.
Time Frame: Baseline, T2 (28-30 weeks post baseline)
Population: The number analyzed includes participants who were able to complete each study visit.
Measure: Mean (Standard Deviation); unit: percent dilation
Arm/Group | Let's Move | Let's Flex
Number analyzed (Participants) | 76 | 39
percent dilation
  Baseline | 4.62 (3.2) | 5.64 (3.8)
  T2 (28-30 weeks post baseline): number analyzed (Participants) | 68 | 33
  T2 (28-30 weeks post baseline) | 4.31 (2.1) | 5.48 (2.6)

19. Other Pre Specified Outcome: Pittsburgh Sleep Quality Index (PSQI) Score
Description: The Pittsburgh Sleep Quality Index (PSQI) is a 19-item measure of the quality and patterns of sleep among adults. Scoring is based on a 0 to 3 Likert scale. The global score is 21; total possible score ranges from 0 to 21. The higher the score the worse the sleep quality.
Time Frame: Baseline, T2 (28-30 weeks post baseline), T3 (56-58 weeks post baseline)
Population: The number analyzed includes participants who were able to complete each study visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Let's Move: Participants in this group will be asked to walk five times per week for twelve weeks for a minimum of 30 minutes in their home while wearing a heart rate monitor and a pedometer. Participants will then enter a maintenance exercise period up to 58 weeks.
  Let's Move Program: Participants will be asked to walk five times per week for twelve weeks for a minimum of 30 minutes while wearing a heart rate monitor and a pedometer. Participants will also receive weekly telephone calls from a member of the research team to monitor walking progress and to change walking duration or intensity level based on their progress.After the twelve week period, participants will enter a maintenance exercise phase for weeks 13-17 in which they will be asked to maintain their exercise regimen.
  Group Motivational Interviewing: Participants will attend four separate group intervention sessions for 2.5 hours for four consecutive weeks at the beginning of the program. Groups will consist of 6-8 members and will focus on the rationale for aerobic exercise, barriers to exercise, finding time for exercise, how to set short and long term exercise goals, and use of self-monitoring to improve exercise engagement.
Arm/Group | Let's Move | Let's Flex
Number analyzed (Participants) | 76 | 39
score on a scale
  Baseline | 7.97 (8.0) | 7.46 (6.0)
  T2 (28-30 weeks post baseline): number analyzed (Participants) | 68 | 33
  T2 (28-30 weeks post baseline) | 7.38 (3.87) | 8.13 (3.87)
  T3 (56-58 weeks post baseline): number analyzed (Participants) | 72 | 31
  T3 (56-58 weeks post baseline) | 7.32 (4.45) | 8.55 (4.45)

20. Other Pre Specified Outcome: Beck Depression Inventory-II (BDI-II) Score
Description: BDI-II is a 21-question multiple-choice self-report inventory, one of the most widely used instruments for measuring the severity of depression. Each answer being scored on a scale value of 0 to 3. Scores range from 0-63. Interpretation: 0 through 9 indicate no or minimal depression; scores from 10 through 18 indicate mild to moderate depression; scores from 19 through 29 indicate moderate to severe depression; and scores from 30 through 63 indicate severe depression.
Time Frame: Baseline, T2 (28-30 weeks post baseline), T3 (56-58 weeks post baseline)
Population: The number analyzed includes participants who were able to complete each study visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Let's Move: Participants will be asked to walk five times per week for twelve weeks for a minimum of 30 minutes while wearing a heart rate monitor and a pedometer. Participants will also receive weekly telephone calls from a member of the research team to monitor walking progress and to change walking duration or intensity level based on their progress.After the twelve week period, participants will enter a maintenance exercise phase for weeks 13-17 in which they will be asked to maintain their exercise regimen.
Arm/Group | Let's Move | Let's Flex
Number analyzed (Participants) | 76 | 39
score on a scale
  Baseline | 6.95 (5.0) | 8.64 (6.0)
  T2 (28-30 weeks post baseline): number analyzed (Participants) | 68 | 33
  T2 (28-30 weeks post baseline) | 8.28 (7.0) | 10.79 (4.0)
  T3 (56-58 weeks post baseline): number analyzed (Participants) | 72 | 31
  T3 (56-58 weeks post baseline) | 7.17 (4.45) | 11.13 (4.45)

21. Other Pre Specified Outcome: Exercise Regimen as Assessed by the Community Healthy Activities Model Program for Seniors (CHAMPS) Questionnaire
Description: The 41-item Community Healthy Activities Model Program for Seniors evaluates weekly duration of various types of physical activity among older adults including light, moderate and vigorous intensity levels. The activity is assessed by hours per week using 6 categories less than 1 hour to 9 or more hours. The values presented below are hours participants indicated they spent in moderate intensity activity levels at the 3 time points over the past 4 weeks. Guidelines suggest 150 minutes (2.5 hours) per week in moderate intensity physical activity, below this number is considered sedentary. We measure change from baseline in time spent in moderate intensity exercise.
Time Frame: Baseline, T2 (28-30 weeks post baseline), T3 (56-58 weeks post baseline)
Population: The number analyzed includes participants who were able to complete each study visit.
Measure: Mean (Standard Deviation); unit: hours per week
Arm/Group | Let's Move | Let's Flex
Number analyzed (Participants) | 76 | 39
hours per week
  Baseline | 9.85 (10.4) | 12.13 (10.4)
  T2 (28-30 weeks post baseline): number analyzed (Participants) | 68 | 33
  T2 (28-30 weeks post baseline) | 12.1 (7.56) | 8.59 (7.56)
  T3 (56-58 weeks post baseline): number analyzed (Participants) | 72 | 31
  T3 (56-58 weeks post baseline) | 9.72 (4.45) | 8.96 (4.45)

22. Other Pre Specified Outcome: V02 Max Rate
Description: V02 max is the maximum rate of oxygen consumption as measured during incremental exercise using the Balke treadmill test. This is an exploratory outcome.
Time Frame: Baseline
Population: Number analyzed includes participants that completed the baseline visit.
Measure: Mean (Standard Deviation); unit: mL/kg/min
Groups:
- Let's Flex Program: Let's Flex Program: Participants will be asked to stretch five times per week for twelve weeks for a minimum of 30 minutes. Participants will also receive weekly telephone calls from a member of the research team to monitor progress and to change duration or intensity level based on their progress. After the twelve week period, participants will enter a maintenance exercise phase for weeks 13-17 in which they will be asked to maintain their exercise regimen.
  Group Motivational Interviewing: Participants will attend four separate group intervention sessions for 2.5 hours for four consecutive weeks at the beginning of the program. Groups will consist of 6-8 members and will focus on the rationale for aerobic exercise, barriers to exercise, finding time for exercise, how to set short and long term exercise goals, and use of self-monitoring to improve exercise engagement.
Arm/Group | Let's Move Program | Let's Flex Program
Number analyzed (Participants) | 76 | 39
mL/kg/min | 20.48 (19.5) | 20.67 (20.3)

23. Other Pre Specified Outcome: Six-minute Walk Test
Description: Measure of functional capacity or submaximal exercise. Scores reflect distance walked in feet for 6 minutes duration. This is an exploratory outcome.
Time Frame: Baseline, T2 (28-30 weeks post baseline), T3 (56-58 weeks post baseline)
Population: The number analyzed includes participants who were able to complete each study visit.
Measure: Mean (Standard Deviation); unit: distance walked in feet
Groups:
- Let's Move: Let's Move Program: Participants will be asked to walk five times per week for twelve weeks for a minimum of 30 minutes while wearing a heart rate monitor and a pedometer. Participants will also receive weekly telephone calls from a member of the research team to monitor walking progress and to change walking duration or intensity level based on their progress.
  After the twelve week period, participants will enter a maintenance exercise phase for weeks 13-17 in which they will be asked to maintain their exercise regimen.
  Group Motivational Interviewing: Participants will attend four separate group intervention sessions for 2.5 hours for four consecutive weeks at the beginning of the program. Groups will consist of 6-8 members and will focus on the rationale for aerobic exercise, barriers to exercise, finding time for exercise, how to set short and long term exercise goals, and use of self-monitoring to improve exercise engagement.
Arm/Group | Let's Move | Let's Flex
Number analyzed (Participants) | 76 | 39
distance walked in feet
  Baseline | 1465.58 (63.58) | 1475.07 (63.58)
  T2 (28-30 weeks post baseline): number analyzed (Participants) | 68 | 33
  T2 (28-30 weeks post baseline) | 1469.3 (261.75) | 1478.11 (261.75)
  T3 (56-58 weeks post baseline): number analyzed (Participants) | 72 | 31
  T3 (56-58 weeks post baseline) | 1497.68 (243.54) | 1475.35 (243.54)

ADVERSE EVENTS:
Time Frame: Patients were followed for the duration of the study (up to 58 weeks post intervention).
Arm/Group | Let's Move Program | Let's Flex Program
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/39
Other Adverse Events (participants affected / at risk) | 0/76 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT02711878/Prot_SAP_001.pdf
  • Informed Consent Form (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT02711878/ICF_000.pdf